CLINICAL TRIAL: NCT04722341
Title: Time-Restricted Eating and Cancer: Clinical Outcomes, Mechanisms, and Moderators
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Alabama at Birmingham (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Sarah Salvy, Professor, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15494; 1R01CA258222-01 (NIH)
Record Dates: First submitted 2020-12-14; First posted 2021-01-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer; Breast Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-Restricted Eating (TRE) (Experimental): 8-hour daily eating period. Participants eating window must start within 2 hours of waking up and no later than 9 am.
  Interventions: Behavioral: Time-Restricted Eating (TRE)
- Control (Active Comparator): More than equal to a 12-hour daily eating period
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Time-Restricted Eating (TRE) — 8-hour daily eating period, starting 1-3 hours after waking up
  Arms: Time-Restricted Eating (TRE)
Behavioral: Control — More than equal to a 12-hour daily eating period
  Arms: Control

SUMMARY:
The purpose of this study is to test whether the timing of meals can improve treatment adverse events, influence tumor biology and alter a person's mood and behaviors.

DETAILED DESCRIPTION:
Combining fasting with chemotherapy is known to cause complete tumor regression and long-term survival in animal models. According to the Differential Stress Sensitization (DSS) theory, acute fasting sensitizes tumor cells to the cytotoxic effects of chemotherapy and radiation, while protecting healthy cells by increasing stress resistance. These effects are believed to be largely mediated via the Insulin-like Growth Factor (IGF-1) pathway. However, extended fasting can be challenging for patients and poses undue health risks. A number of alternative intermittent fasting regimens have been proposed to overcome the challenges of prolonged caloric restriction. One promising approach is time-restricted eating (TRE), which involves eating within a period of 10 hours or less, followed by fasting for at least 14 hours daily. TRE does not involve extended caloric restriction, and because of its simplicity, it may be more sustainable than other fasting regimens. TRE improves several cardiometabolic endpoints independent of calorie restriction in both animals and humans, including insulin sensitivity, blood pressure, fat oxidation, and hunger. Our team's pilot and feasibility trials suggest that TRE may also have anti-cancer effects: it decreases IGF-1 levels, reduces oxidative stress, upregulates antioxidant defenses, and enhances autophagy. Moreover, our data suggest TRE is sustainable, as participants were adherent 6.0 plus or minus 0.8 days/week over a 14-week period. These findings lead to the following provocative question: Can TRE reduce treatment-related toxicity, induce tumor regression, and improve both patient-reported and clinical outcomes? We propose to conduct the largest randomized controlled trial of any form of intermittent fasting in patients undergoing cancer treatment. We focus on patients with localized rectal or breast cancer because it is one of the few treatment paradigms in which tumor characteristics can be measured before and after chemoradiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Any sex/gender of any ethnic/racial background
* Age greater than or equal to 18 years
* Histologically-confirmed rectal cancer stage II, III, or IV (if curative) or human epidermal growth factor receptor 2-positive (HER2+) or triple negative breast cancer stage I, II, or III (only if definitive intent) per American Joint Committee on Cancer (AJCC) criteria
* BMI 18.5 kg/m2 or greater
* Receiving either neoadjuvant therapy with curative intent (breast cancer patients) or total neoadjuvant therapy with a 5-fluorouracil-based regimen and curative intent (rectal cancer patients)
* Has completed ≤ 4 weeks of neoadjuvant treatment prior to study enrollment
* Willing and able to adhere to the assessments, visit schedules, prohibitions, and restrictions

Exclusion Criteria:

* History of cytotoxic chemotherapy less than or equal to 12 months prior to rectal or breast cancer diagnosis
* Allergic reaction to any of the treatment agents
* Any prior pelvic radiotherapy
* Currently active second malignancy other than non-melanoma skin cancers or cervical carcinoma in situ
* History of GI perforation ≤12 months prior to enrollment
* History of predisposing colonic or small bowel disorders with severe or rapidly worsening symptoms (not related to current cancer symptoms)
* Receiving any parenteral nutrition or enteral (tube) feeding or using similar nutritional supplement during the study period
* History of uncontrolled congestive heart failure defined as ew York Heart Association Class (NYHA) Class III or greater
* Pre-existing grade ≥3 neuropathy
* Currently participating in or has participated in a study of an investigational agent or investigational device ≤4 weeks of the first dose of treatment
* Pregnant or breastfeeding
* Currently perform overnight shift work more than one day/week on average
* Strictly adhering to a <10-hour eating window on most days
* Known psychiatric or substance abuse disorders that would interfere with adhering to the requirements of the trial
* Medical condition or laboratory abnormality that could impact participant safety or data validity, in the opinion of the medical investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) and Organ Preservation Rate | at end of 6-month intervention
  Measures whether participants achieve either a pathologic complete response (no invasive cancer is found in the removed tumor or sampled lymph nodes) or organ preservation at the end of treatment. For rectal cancer, organ preservation is defined as a complete or near-complete clinical response after therapy that allows the patient to safely avoid surgery, based on findings from exam, endoscopy, and MRI. Quantified as a percentage (%).
Patient-Reported AEs (PRO-CTCAEs) | at end of 6-month intervention
  Adverse events as measured by the PRO-CTCAE (version 5), which includes about three dozen toxicities that patients can systematically document the frequency, severity (and interference of each toxicity).

SECONDARY OUTCOMES:
Clinical Response | at end of 6-month intervention
  Clinical response at end of treatment, categorized as: complete (no detectable disease on exam, endoscopy, or MRI); near-complete (minimal residual abnormality); partial (≥30% tumor decrease); stable disease; or progressive disease (≥20% tumor increase). We will also report the objective response rate (complete + near-complete + partial), percent with complete/near-complete responses, and percent with progressive disease. For breast cancer, responses may be estimated by physicians or MRI technicians. Values will also be expressed as percentages.
Tumor Response | at end of 6 month intervention
  Different scales by cancer type. Rectal cancer, using MRI Tumor Regression Grade (1-5, with 1 = complete response) at end of treatment and the Neoadjuvant Rectal (NAR) score (0-100) at baseline and post-intervention. Breast cancer measured using the Residual Cancer Burden (RCB) score (0-4), where 0 indicates a pathologic complete response.
Provider-Reported AEs (Treatment Related Toxicities) | at end of 6 month intervention
  Measures treatment-related adverse events (AEs) reported by providers from the start of therapy to the day before surgery. AEs are graded using CTCAE v5, and we will report totals as well as Grade 1-2 and Grade 3-4 events. The Toxicity Index (TI) will also be calculated, which ranges from 0 to 5.83.
Health-Related Quality of Life | at end of 6 month intervention
  Assessed at each testing visit using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core 30 (EORTC QLQ-C30) for all participants, the QLQ-breast cancer 23 (QLQ-BR32) for breast cancer, and the QLQ-rectal cancer 29 (QLQ-CR29) for rectal cancer. All scales are scored from 0-100, with higher functional and global health scores indicating better quality of life and higher symptom scores indicating worse symptoms. The QLQ-C30 includes five functional scales, three symptom scales, and a global quality-of-life scale, while the BR23 and CR29 include cancer-specific functional and symptom scales.

OTHER OUTCOMES:
Complete Blood Counts (CBCs) | at end of 6 month intervention
  Obtained through each site's hospital laboratory; results from within two weeks of a testing visit may be used instead of a new draw. All CBC values collected from consent to surgery will be included in analyses. For rectal cancer patients, Carcinoembryonic Antigen (CEA) and Carbohydrate Antigen 19-9 (CA 19-9) results from consent to surgery will also be extracted from the medical record.
Protein Expression Related to Cell Growth and Death | at end of 6 month intervention
  Measure molecular markers representing cell growth and death and stress resistance, including Antigen Kiel 67 (Ki-67; cell proliferation), caspase 3 (apoptosis), microtubule-associated protein light chain 3B (LC3-I/LC3-II; autophagy), and phosphorylated histone H2AX (γ-H2AX; DNA damage). Protein expression will be measured in formalin-fixed paraffin-embedded tumor and adjacent normal tissue obtained from both biopsy (baseline) and surgical resection (post-intervention). Values will be expressed as fold changes.
Total Antioxidant Capacity | at end of 6 month intervention
  Measured in serum and/or peripheral blood mononuclear cells (PBMCs) collected at each testing visit. PBMCs isolated from whole blood. Values expressed in A.U.
Body weight | at end of 6 month intervention
  Measured at each in-person visit after ≥8 hours of fasting, using a calibrated metabolic scale. Interim non-fasting weights will be extracted from the medical record when available. Weight will be recorded in kilograms to the nearest 0.1 kg.
Blood pressure | at end of 6 month intervention
  Systolic and diastolic blood pressure will be measured using an automated blood pressure monitor following American Heart Association/American College of Cardiology guidelines. After a five-minute seated rest, three readings will be taken 1-2 minutes apart; the average of the two closest values will be used. If blood pressure cannot be collected at a testing visit, values from the nearest clinical encounter will be extracted from the medical record. Blood pressure is reported in mm Hg.
Heart Rate | at end of 6 month intervention
  Measured concurrently with blood pressure using the automated monitor. Three readings will be obtained after a five-minute rest, and the average of the two closest measurements will be used. Heart rate is recorded in beats per minute (bpm).
Adherence | at end of 6 month intervention
  Self-reported in weekly surveys, with participants recording daily eating start/stop times and reasons for non-adherence using surveys. Quantified as the percentage of adherent days (eating window followed within 30 minutes; missing days counted as non-adherent) and the median eating duration.
Fatigue | at end of 6 month study
  Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS®) Fatigue subscale. Items are rated on a Likert scale and converted to T-scores (mean = 50, standard deviation (SD) = 10), with higher scores indicating greater fatigue.
Social Functioning | at end of 6 month study
  Measured using:
  * University of California at Los Angeles (UCLA) 3-Item Loneliness Scale: scores range from 3-9, with higher scores indicating greater loneliness.
  * PROMIS® Satisfaction with Participation in Discretionary Social Activities (Short Form 7a): Likert-scale items converted to T-scores (mean = 50, SD = 10), with higher scores indicating greater social satisfaction.
Physical Functioning | at end of 6 month study
  Assessed using the PROMIS® Physical Function subscale (Likert-scale items). Scores are converted to T-scores (mean = 50, SD = 10), with higher scores indicating better physical function.
Mood | at end of 6 month study
  Assessed using the PROMIS® Anxiety subscale. Responses are scored on Likert-scale items and converted to age-standardized T-scores (mean = 50, SD = 10), with higher scores indicating greater anxiety.
Dietary Intake | at end of 6 month intervention
  Assessed using three-day food records (two weekdays and one weekend day) in conjunction with each testing visit. Measures will include total energy intake, Healthy Eating Index (HEI-2015) scores, and intake of key dietary components such as added sugar, fruits and vegetables, solid fats, alcohol, sodium, and fats.
Appetite | at end of 6 month intervention
  Assessed using two self-report scales: (1) a retrospective 5-point Likert scale rating the frequency of hunger and fullness over the past week, and (2) a 100-point visual analog scale (0 = "Not at all," 100 = "Extremely") rating typical hunger and fullness levels during eating and fasting windows.
Eating Behavior | at end of 6 month intervention
  Assessed using the Dutch Eating Behavior Questionnaire (DEBQ), which measures three domains: emotional eating, external eating, and restrained eating. Scores reflect the frequency of behaviors within each domain, with higher scores indicating greater endorsement of that eating pattern.
Physical Activity | at end of 6 month intervention
  Assessed using an ActiGraph GT9X accelerometer. Activity outcomes derived using GGIR algorithms, including metabolic equivalents (METs) and the percentage of time spent in sedentary, light, moderate, and vigorous activity (Friedson algorithms). Self-reported physical activity measured using the General Physical Activity Questionnaire (GPAQ), MET-minutes per week for moderate and vigorous activity and estimates daily sedentary time.
Sleep | at end of 6 month intervention
  Measured using accelerometer-derived estimates from the ActiGraph GT9X (processed with GGIR) for sleep duration, timing, and sleep efficiency. Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI; global score 0-21, with higher scores indicating poorer sleep), and sleep duration and timing will be self-reported using the Munich Chronotype Questionnaire (MCTQ). Values for the latter will be reported in either minutes or hours.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, West Hollywood, California

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT04722341/Prot_SAP_000.pdf